CLINICAL TRIAL: NCT05012943
Title: A Randomized, Observer-Blind, Controlled Study to Assess the Safety, Immunogenicity and Efficacy of the SARS-CoV-2 Self- Amplifying RNA Vaccine ARCT-154 in Adults
Brief Title: The ARCT-154 Self-Amplifying RNA Vaccine Efficacy Study (ARCT-154-01)
Acronym: ARCT-154-01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vinbiocare Biotechnology Joint Stock Company (Industry)
Collaborators: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ARCT-154-01
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: COVID-19 Vaccines
Keywords: ARCT-154; COVID-19; SARS-CoV-2; Immunogenicity; Efficacy
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Phase 1, 2, 3a, 3b: Participants will be randomly assigned to a study group that will receive up to 2 vaccination series. Each vaccination series comprises two vaccinations at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series at around 2 months after the first series on Day 92 and 120. Each participant is planned to receive a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series.
  Participants in Phase 2, 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series will be rerandomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120.
  Phase 3c: Participants will be randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Observer-blind design:
  Investigators, site staff, participants, CRO staff, Sponsor representatives with oversight of study conduct or study-related assessments will remain blinded to vaccine assignments for the study duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- ARCT-154 (Experimental): Each participant is planned to receive a two-dose vaccination series of ARCT-154 at a dose of 5 µg with 28 day interval in the first vaccination series.
  Interventions: Biological: ARCT-154 Self-Amplifying RNA SARS-CoV-2 Vaccine
- Placebo (Placebo Comparator): Each participant is planned to receive a two-dose vaccination series of placebo (normal saline) with 28 day interval in the first vaccination series.
  Interventions: Other: Placebo (normal saline)
- Astra Zeneca COVID-19 vaccine (Active Comparator): Each participant is planned to receive a two-dose vaccination series of Astra Zeneca COVID-19 vaccine with 28 day interval in the first vaccination series.
  Interventions: Biological: Astra Zeneca COVID-19 vaccine

INTERVENTIONS:
Biological: ARCT-154 Self-Amplifying RNA SARS-CoV-2 Vaccine — ARCT-154 Self-Amplifying RNA SARS-CoV-2 Vaccine
  Arms: ARCT-154
Other: Placebo (normal saline) — Normal saline with the same volume as of ARCT-154
  Arms: Placebo
Biological: Astra Zeneca COVID-19 vaccine — Astra Zeneca COVID-19 vaccine (ChAdOx1 nCoV-19)
  Arms: Astra Zeneca COVID-19 vaccine

SUMMARY:
This is a Phase 1/2/3, randomized, placebo-controlled, observer-blind study designed to evaluate the safety, immunogenicity and efficacy of ARCT-154 in adult participants to be enrolled in Vietnam.

This study consists of four parts:

Part 1 (Phase 1) will evaluate the safety of the study vaccines in 100 healthy individuals.

Part 2 (Phase 2) will evaluate the safety and immunogenicity of the study vaccines in 300 healthy individuals.

Part 3 (Phase 3a) will evaluate the safety, immunogenicity, and efficacy of the study vaccines in 600 individuals with and without underlying medical conditions.

Part 4 (Phase 3b) will evaluate the safety and efficacy of the study vaccines in 16,000 individuals with and without underlying medical conditions.

Part 5 (Phase 3c) will evaluate the safety and non-inferiority in immunogenicity of ARCT-154 vaccine vs. Astra Zeneca COVID-19 vaccine (ChAdOx1 nCoV-19) in 2400 individuals with and without underlying medical conditions.

In Phase 1, healthy individuals 18 to < 60 years of age will be enrolled. In Phase 2, 3a, and 3b, individuals 18 years of age and older will be enrolled including individuals with underlying medical conditions that put them at higher risk of complications of COVID-19 disease.

Phase 1, Phase 2, Phase 3a and Phase 3b participants will be randomly assigned to a study group that will receive up to 2 vaccination series. Each vaccination series comprises two vaccinations at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series around 2 months after the first series (on Day 92 and 120).

Participants of Phase 2, 3a who received 2 doses of ARCT-154 vaccine will be rerandomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120.

For Phase 1, Phase 3b and participants in Phase 2 and 3a that received placebo in the first vaccination series, the participants will be switched over to the opposite vaccine in the second series.

There is no second vaccination series for Phase 3c as all participants receive active vaccine in the initial series.

DETAILED DESCRIPTION:
Phase 1 will enroll 100 healthy participants that are randomly assigned 3:1 to receive ARCT-154 or placebo (75:25) for the initial series of vaccinations.

In Phase 2, 300 participants will be randomly assigned 3:1 to receive ARCT-154 or placebo for the initial series of vaccinations. Participants that received ARCT-154 in the initial series will be rerandomized 3:1 to receive ARCT or placebo on Day 92 followed by placebo on Day 120.

In Phase 3a, 600 participants will be randomly assigned 3:1 to receive ARCT-154 or placebo for the initial series of vaccinations. Participants that received ARCT-154 in the initial series will be rerandomized 3:1 to receive ARCT or placebo on Day 92 followed by placebo on Day 120.

In Phase 3b, ~16,000 participants will be randomly assigned 1:1 to receive ARCT-154 or placebo for the initial series of vaccinations.

In Phase 3c, ~2,400 participants will be randomly assigned 1:1 to receive ARCT-154 or Astra Zeneca COVID-19 vaccine. Blood samples will be collected and reserved for Immunogenicity evaluation for the first 1500 participants (3c-1) and assays for immunogenicity evaluation will be performed for the first 800 participants.

Phase 1 participants must be <60 years of age and healthy. Phase 2, 3a, and 3b and 3c participants will include elderly (≥60 years) and those with comorbidities.

For Phase 2, 3a, 3b and 3c, prior to randomization, participants will be stratified by age (< 60 or ≥ 60 years of age) and for participants < 60 years of age by risk of severe COVID 19. Participants will be followed up for approximately 1 year after completion of the initial vaccination series.

An independent Data and Safety Monitoring Board (DSMB) will perform ongoing review of blinded and unblinded data.

An independent blinded adjudication committee will adjudicate all suspected COVID-19 cases to determine if they meet the primary endpoint requirements.

ELIGIBILITY:
Inclusion Criteria:

Individuals who:

1. are able to provide consent
2. agree to comply with all study visits and procedures
3. are of childbearing potential and sexually active must be willing to adhere to contraceptive requirements
4. are male or female ≥18 years of age (or, for Phase 1, 18 to < 60 years of age)
5. are at higher risk of developing COVID-19 based on where they work or live

Exclusion Criteria:

Individuals who:

1. Significant infection or other acute illness, including body temperature >100.4°F (>38.0°C) on the day prior to or Day 1. Participants meeting this criterion may be rescheduled within the relevant window periods. Afebrile participants with minor illnesses can be enrolled at the discretion of the investigator.
2. Pregnant or breastfeeding.
3. Known history of COVID-19 (asymptomatic SARS-CoV-2 infection and/or nucleocapsid positive test is not exclusionary).
4. Close contact with a person known to be SARS-CoV-2 positive or with a clinical diagnosis of COVID-19 within 7 days prior to enrollment. Participants meeting this criterion who remain asymptomatic for 7 days may be rescheduled for enrollment within the relevant windows.
5. Known history of anaphylaxis, urticaria, or other significant adverse reaction to the vaccine or its excipients.
6. Known history of anaphylaxis to other vaccines.
7. Bleeding disorder considered a contraindication to intramuscular (IM) injection or phlebotomy.
8. Immunosuppressive or immunodeficient state, asplenia, recurrent severe infections, or known to be HIV positive.
9. An underlying clinically significant acute or chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

   Prior/Concomitant Therapy
10. Has previously received investigational or approved MERS-CoV, SARS-CoV, SARS-CoV-2 vaccines or who have plans to receive off-study COVID-19 vaccines.
11. Has received a live replicating vaccine within 28 days prior to each study vaccination or a licensed inactivated or non-replicating vaccine within 14 days prior to first study vaccination.
12. Has received treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, within 6 months prior to Screening, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days prior to first study vaccine administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
13. Has received systemic immunoglobulins or blood products within 3 months prior to first study vaccine administration or plans to receive such products during the study.

    Other Exclusions
14. Demonstrated inability to comply with the study procedures.
15. Investigator site staff members, employees of the Sponsor or the CRO directly involved in the conduct of the study, or site staff members otherwise supervised by the investigator, or immediate family members of any of the previously mentioned individuals.
16. Other restrictions apply to Phase 1 participants to ensure they are healthy.

Additional Exclusion Criteria for Phase 3c Participants Only:

No contraindications (as specified in the prescribing information) to receiving the ChAdOx1 vaccine.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19474 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Vietnam (3):
  - Hanoi Medical University, Hanoi, Hanoi
  - Military Medical University, Hanoi, Hanoi
  - Pasteur Institute, Ho Chi Minh City, Ho Chi Minh

IPD SHARING:
Plan to Share IPD: No
IPD is the sole property of VinBioCare. VinBioCare may share a copy of the study IPD with their collaborative partners if requested.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As pre-specified, data were collected and are reported per vaccine group overall for all study phases combined. Data are reported per first treatment received.
Groups:
- Placebo: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 micrograms (µg) or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per initial treatment received. Data in this arm are presented pooled for participants who initially received placebo in Phases 1, 2, 3a, 3b.
- ARCT-154: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series (Day 1 and Day 29) of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per initial treatment received. Data in this arm are presented pooled for participants who initially received ARCT-154 in Phases 1, 2, 3a, 3b, 3c.
- Astra Zeneca COVID-19 vaccine: Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]) on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for Astra Zeneca COVID-19 vaccine received in Phase 3c.
Period: Overall Study
Arm/Group | Placebo | ARCT-154 | Astra Zeneca COVID-19 vaccine
Started | 8300 | 9992 | 1182
Phase 1: Received ARCT-154 D1-92 | 0 | 74 | 0
Phase 1: Received Placebo D1-92 | 26 | 0 | 0
Phase 1: Received Initially Placebo, ARCT-154 D92-EOS | 23 | 0 | 0
Phase 1: Received Initially ARCT-154, Placebo D92-EOS | 0 | 67 | 0
Phase 3b: Received ARCT-154 D1-92 | 0 | 8059 | 0
Phase 3b: Received Placebo D1-92 | 8041 | 0 | 0
Phase 3b: Received Initially Placebo, ARCT-154 D92-EOS | 7350 | 0 | 0
Phase 3b: Received Initially ARCT-154, Placebo D92-EOS | 0 | 7458 | 0
Phase 2: Received ARCT-154 D1-92 | 0 | 226 | 0
Phase 2: Received Placebo D1-92 | 75 | 0 | 0
Phase 3a: Received ARCT-154 D1-92 | 0 | 448 | 0
Phase 3a: Received Placebo D1-92 | 152 | 0 | 0
Phase 2 Received Initially Placebo, ARCT-154 D92-EOS | 72 | 0 | 0
Phase 2 Received Initially ARCT-154, Placebo D92-EOS | 0 | 55 | 0
Phase 3a Received Initially Placebo, ARCT-154 D92-EOS | 137 | 0 | 0
Phase 3a Received Initially ARCT-154, Placebo D92-EOS | 0 | 98 | 0
Phase 3C: Received ARCT-154 | 0 | 1186 | 0
Phase 2 Received Initially ARCT-154, ARCT-154 D92-EOS | 0 | 159 | 0
Phase 3a Received initially ARCT-154, ARCT-154 D92-EOS | 0 | 324 | 0
Completed | 7207 | 8942 | 1155
Not Completed | 1093 | 1050 | 27
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Withdrawal by Subject | 1052 | 1006 | 20
Not completed — Death | 25 | 17 | 4
Not completed — Lost to Follow-up | 11 | 24 | 3
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Other than Specified | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, which included all participants who received any dose of study vaccine (ARCT-154 or placebo or ChAdOx1). As pre-specified, data were collected and are reported according to the initial study vaccine received, pooled per treatment received for Phase 1/2/3a/3b (ARCT-154/placebo), and separately for ChAdOx1 and ARCT-154 for Phase 3c. Participants are counted only once, baseline data were collected and are reported based on initial treatment received.
Groups:
- ARCT-154: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series (Day 1 and Day 29) of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for ARCT-154 received in Phases 1, 2, 3a, 3b.
- Placebo: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 micrograms (µg) or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for placebo received in Phases 1, 2, 3a, 3b.
- Phase 3c: ARCT-154: Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover). Data in this arm are presented pooled for ARCT-154 vaccine received in Phase 3c.
- Total: Total of all reporting groups
Arm/Group | ARCT-154 | Placebo | Phase 3c: ARCT-154 | Astra Zeneca COVID-19 vaccine | Total
Number analyzed (Participants) | 8807 | 8294 | 1186 | 1180 | 19467
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 47.0 [37.0 to 57.0] | 48.0 [37.0 to 57.0] | 52.0 [42.0 to 61.0] | 52.0 [41.0 to 61.0] | 48.0 [37.0 to 57.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4441 | 4206 | 603 | 613 | 9863
  Male | 4366 | 4088 | 583 | 567 | 9604
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  The Kinh | 8757 | 8239 | 1185 | 1177 | 19358
  Other | 50 | 55 | 1 | 3 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Local Adverse Reactions (ARs)
Description: Solicited local ARs included injection site erythema, injection site pain, injection site induration/swelling, and injection site tenderness. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Within 7 days after Dose 1 and Dose 2 (up to Day 7 and 36)
Population: Reactogenicity Analysis Set, all participants who received any dose of study vaccine (ARCT-154 or placebo or ChAdOx1) and provided at least 1 reactogenicity diary report. As pre-specified, data are presented pooled per treatment received for Phase 1/2/3a/3b, and separately for ARCT-154 for Phase 3c. Overall number of participants analyzed = number of participants evaluable for the endpoint. Number analyzed = number of participants with evaluable data at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo | Phase 3c: ARCT-154 | Astra Zeneca COVID-19 vaccine
Number analyzed (Participants) | 8688 | 8151 | 1182 | 1180
Participants
  Dose 1: number analyzed (Participants) | 8688 | 8151 | 1182 | 1176
  Dose 1 | 4060 | 909 | 467 | 416
  Dose 2: number analyzed (Participants) | 8459 | 7915 | 1150 | 1149
  Dose 2 | 2852 | 612 | 286 | 183

2. Primary Outcome: Number of Participants Reporting Solicited Systemic ARs
Description: Solicited systemic ARs included arthralgia, chills, diarrhea, dizziness, fatigue, fever (categorized by measured body temperature), headache, myalgia, and nausea/vomiting. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Within 7 days after Dose 1 and Dose 2 (up to Day 7 and 36)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo | Phase 3c: ARCT-154 | Astra Zeneca COVID-19 vaccine
Number analyzed (Participants) | 8688 | 8151 | 1182 | 1180
Participants
  Dose 1: number analyzed (Participants) | 8688 | 8151 | 1182 | 1176
  Dose 1 | 4375 | 2620 | 638 | 657
  Dose 2: number analyzed (Participants) | 8459 | 7915 | 1150 | 1149
  Dose 2 | 3718 | 1889 | 477 | 331

3. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AEs were defined as any spontaneously reported or discovered AE. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Approximately 28 days after Dose 1 and Dose 2 (Day 1 to Day 29 and Day 29 to Day 57)
Population: Safety Analysis Set, all participants who received any dose of study vaccine (ARCT-154 or placebo or ChAdOx1). Participants were analyzed according to the study vaccine received. As pre-specified, data are presented pooled per treatment received for Phase 1/2/3a/3b, and separately for ARCT-154 for Phase 3c. Overall number of participants analyzed = number of participants evaluable for the endpoint. Number analyzed = number of participants with evaluable data at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo | Phase 3c: ARCT-154 | Astra Zeneca COVID-19 vaccine
Number analyzed (Participants) | 8807 | 8294 | 1186 | 1180
Participants
  Dose 1 | 1323 | 1198 | 260 | 252
  Dose 2: number analyzed (Participants) | 8599 | 8067 | 1171 | 1167
  Dose 2 | 1232 | 1311 | 226 | 225

4. Primary Outcome: Number of Participants Reporting Medically Attended Adverse Events (MAAEs), Serious Adverse Events (SAEs) and AEs Leading to Discontinuation
Description: An MAAE was defined as an AE that led to an unscheduled visit (including a telemedicine visit) with a healthcare provider ([HCP], e.g., nurse, nurse practitioner, physician's assistant, physician). An SAE was defined as any event that resulted in death, was immediately life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or was a congenital anomaly/birth defect arising from a pregnancy conceived after receipt of study vaccine. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 to Day 92
Population: Safety Analysis Set, all participants who received any dose of study vaccine (ARCT-154 or placebo or ChAdOx1). Participants were analyzed according to the study vaccine received. As pre-specified, data are presented pooled per treatment received for Phase 1/2/3a/3b, and separately for ARCT-154 for Phase 3c. Overall number of participants analyzed = number of participants evaluable for the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo | Phase 3c: ARCT-154 | Astra Zeneca COVID-19 vaccine
Number analyzed (Participants) | 8807 | 8294 | 1186 | 1180
Participants
  MAAEs | 1132 | 1284 | 148 | 146
  SAEs | 133 | 217 | 22 | 35
  AEs Leading to Discontinuation | 6 | 18 | 0 | 1

5. Primary Outcome: Number of Participants With Neutralizing Antibody (NAb) Responses
Description: Data are presented for the number of participants with a NAb seroconversion response as determined by the surrogate virus neutralization test (sVNT). Seroconversion was defined as a ≥4-fold increase in antibody concentration from baseline.
Time Frame: Day 57
Population: Immunogenicity Analysis Set, all participants who received all protocol required doses of vaccine up to evaluation timepoint, no evidence of prior severe acute respiratory syndrome coronavirus 2(SARS-CoV-2) infection at Day 1, at least 1 valid post-vaccination immunogenicity assay result. As pre-specified, data is pooled per treatment received for participants in Phase 1, 2, 3a. Overall number of participants analyzed=number of participants evaluable for the endpoint at the specified timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- ARCT-154: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series (Day 1 and Day 29) of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for ARCT-154 received in Phases 1, 2, 3a.
- Placebo: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 micrograms (µg) or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for placebo received in Phases 1, 2, 3a.
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 699 | 231
Participants | 658 | 1

6. Primary Outcome: Number of Participants With a First Occurrence of Coronavirus Disease 2019 (COVID-19)
Description: COVID-19 was defined as a positive SARS-CoV-2 test and at least one of the following that was a new or worsening finding: ⦁ Fever or chills ⦁ Cough ⦁ Shortness of breath or difficulty breathing ⦁ Fatigue ⦁ Muscle or body aches ⦁ Headache ⦁ New loss of taste or smell ⦁ Sore throat ⦁ Congestion or runny nose ⦁ Nausea or vomiting ⦁ Diarrhea Data are presented for the number of participants with a first occurrence of COVID-19 with no evidence of prior infection.
Time Frame: Day 36 to Day 92
Population: Modified Intent-to-Treat (mITT) Analysis Set (Phase 3b), which included all participants who received all protocol-required doses of study vaccine up to the evaluation timepoint concerned, and who had no evidence of SARS-CoV-2 infection on Day 1 or up to 7 days after the 2nd study vaccination. As pre-specified, data are presented pooled per treatment received and for participants in Phase 3b only. Number of participants analyzed = those with evaluable data for this endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- ARCT-154: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series (Day 1 and Day 29) of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for ARCT-154 received in Phase 3b.
- Placebo: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 micrograms (µg) or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for placebo received in Phase 3b.
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 7762 | 7696
Participants | 200 | 440

7. Secondary Outcome: Geometric Mean Titers of SARS-CoV-2 Neutralizing Antibodies
Time Frame: Days 1, 29, 57 and 92
Population: Immunogenicity Analysis Set, all participants who received all protocol required doses of study vaccine up to evaluation timepoint, no evidence of prior SARS-CoV-2 infection at Day 1, with at least 1 valid post-vaccination immunogenicity assay result. As pre-specified, data is pooled per treatment received for participants in Phase 1, 2, 3a. Overall number of participants analyzed=participants evaluable for endpoint. Number analyzed=participants with evaluable data at the specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 724 | 242
IU/mL
  Day 1 | 15.3 [15.2 to 15.4] | 15.2 [15.0 to 15.3]
  Day 29: number analyzed (Participants) | 719 | 240
  Day 29 | 60.7 [56.6 to 65.1] | 15.7 [15.2 to 16.1]
  Day 57: number analyzed (Participants) | 700 | 231
  Day 57 | 221.4 [207.6 to 236.1] | 15.2 [15.2 to 15.2]
  Day 92: number analyzed (Participants) | 668 | 221
  Day 92 | 209.6 [188.2 to 233.3] | 20.3 [18.0 to 22.9]

8. Secondary Outcome: Geometric Mean Fold Rise in SARS-CoV-2 Neutralizing Antibody Titers
Time Frame: Days 29, 57, 92
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 718 | 240
Ratio
  Day 29 | 4.0 [3.7 to 4.3] | 1.0 [1.0 to 1.1]
  Day 57: number analyzed (Participants) | 699 | 231
  Day 57 | 14.5 [13.6 to 15.5] | 1.0 [1.0 to 1.0]
  Day 92: number analyzed (Participants) | 667 | 221
  Day 92 | 13.7 [12.3 to 15.3] | 1.3 [1.2 to 1.5]

9. Secondary Outcome: Number of Participants Seroconverting for Neutralizing Antibodies
Description: Seroconversion was defined as a ≥4-fold increase in antibody concentration from baseline as measured by the sVNT test. Data are presented for the number of participants seroconverting for neutralizing antibodies.
Time Frame: Days 29, 57 and 92
Population: Immunogenicity Analysis Set, all participants who received all protocol required doses of study vaccine up to evaluation timepoint, no evidence of prior SARS-CoV-2 infection at Day 1, with at least 1 valid post-vaccination immunogenicity assay result. As pre-specified, data is pooled per treatment received for participants in Phase 1, 2, 3a. Overall number of participants analyzed=participants evaluable for the endpoint. Number analyzed=participants with evaluable data at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 718 | 240
Participants
  Day 29 | 388 | 4
  Day 57: number analyzed (Participants) | 699 | 231
  Day 57 | 658 | 1
  Day 92: number analyzed (Participants) | 667 | 221
  Day 92 | 571 | 21

10. Secondary Outcome: Geometric Mean Concentration of Spike Protein Immunoglobulin G (IgG) Binding Antibodies
Time Frame: Days 1, 29, 57, 92
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: units (U)/ milliliter (mL)
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 725 | 242
units (U)/ milliliter (mL)
  Day 1 | 0.3 [0.3 to 0.3] | 0.3 [0.3 to 0.3]
  Day 29: number analyzed (Participants) | 719 | 240
  Day 29 | 2.1 [2.0 to 2.3] | 0.3 [0.3 to 0.3]
  Day 57: number analyzed (Participants) | 701 | 231
  Day 57 | 20.3 [19.0 to 21.7] | 0.3 [0.3 to 0.3]
  Day 92: number analyzed (Participants) | 668 | 221
  Day 92 | 11.9 [10.6 to 13.3] | 0.4 [0.3 to 0.5]

11. Secondary Outcome: Geometric Mean Fold Ratio of Spike Protein IgG Binding Antibodies
Time Frame: Days 29, 57, 92
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 719 | 240
ratio
  Day 29 | 7.5 [6.9 to 8.1] | 1.0 [0.9 to 1.0]
  Day 57: number analyzed (Participants) | 701 | 231
  Day 57 | 71.4 [66.6 to 76.5] | 1.0 [0.9 to 1.0]
  Day 92: number analyzed (Participants) | 668 | 221
  Day 92 | 42.0 [37.5 to 47.1] | 1.5 [1.2 to 1.8]

12. Secondary Outcome: Number of Participants Seroconverting for Spike Protein IgG Binding Antibodies
Description: Seroconversion was defined as a ≥4-fold increase in antibody concentration from baseline. Data are presented for the number of participants seroconverting for spike protein IgG binding antibodies.
Time Frame: Days 29, 57, 92
Population: Immunogenicity Analysis Set, all participants who received all protocol-required doses of study vaccine up to evaluation timepoint, no evidence of prior SARS-CoV-2 infection at Day 1, with at least 1 valid post-vaccination immunogenicity assay result. As pre-specified, data is pooled per treatment received for participants in Phase 1, 2, 3a. Overall number of participants analyzed=participants evaluable for the endpoint. Number analyzed=participants with evaluable data at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 719 | 240
Participants
  Day 29 | 527 | 3
  Day 57: number analyzed (Participants) | 701 | 231
  Day 57 | 698 | 3
  Day 92: number analyzed (Participants) | 668 | 221
  Day 92 | 652 | 29

13. Secondary Outcome: Number of Participants Seroconverting on Neutralizing Antibody Responses by Plaque Reduction Neutralization Test at 50% Reduction (PRNT50)
Description: The plaque reduction neutralization test (PRNT) is a live virus assay. Neutralizing antibody titers were calculated as the highest serum dilution that resulted in 50% reduction in the number of virus plaques (PRNT50). Data presented is for the ancestral-clinical isolate variant. Data are presented for the number of participants that demonstrated seroconversion (as defined by 4-fold increase in neutralizing antibody concentration from baseline) on PRNT50.
Time Frame: Days 29 and 57
Population: Immunogenicity Analysis Set, all participants who received all protocol-required doses of study vaccine up to evaluation timepoint, no evidence of prior SARS-CoV-2 infection at Day 1, with at least 1 valid post-vaccination immunogenicity assay result. As pre-specified, data is pooled per treatment received for participants in Phases 1 and 2. Overall number of participants analyzed=participants evaluable for the endpoint. Number analyzed=participants with evaluable data at specified timepoints.
Measure: Count of Participants; unit: Participants
Groups:
- ARCT-154: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series (Day 1 and Day 29) of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for ARCT-154 received in Phases 1 and 2.
- Placebo: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 micrograms (µg) or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for placebo received in Phases 1 and 2.
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 111 | 37
Participants
  Day 29 | 17 | 0
  Day 57 | 86 | 0

14. Secondary Outcome: Number of Participants With a First Occurrence of Severe COVID-19
Description: Number of participants with a first occurrence of severe COVID-19 in participants with no evidence of prior infection. Severe COVID-19 was defined as a positive SARS-CoV-2 test, symptoms per protocol-defined COVID-19 and any of the following: Clinical signs at rest indicative of severe systemic illness: - Respiratory rate ≥30 per minute, - Heart rate ≥125 per minute, - Oxygen saturation (SpO2) ≤93% on room air at sea level or partial pressure of oxygen (PO2)/fraction of inspired oxygen (FiO2) <300 millimeter of mercury (mm Hg) - Respiratory failure (defined as needing high flow oxygen, noninvasive ventilation, mechanical ventilation or extracorporeal membrane oxygenation [ECMO]); Evidence of shock: - Systolic blood pressure (SBP) <90 mm Hg, or - Diastolic blood pressure (DBP) <60 mm Hg, or requiring vasopressors, - Significant acute renal, hepatic, or neurologic dysfunction - Admission to an intensive care unit (ICU) - Death
Time Frame: Day 36 to Day 92
Population: Modified Intent-to-Treat (mITT) Analysis Set (pooled for Phases 1/2/3a/3b), which included all participants who received all protocol-required doses of study vaccine up to the evaluation timepoint concerned, and who had no evidence of SARS-CoV-2 infection on Day 1 or up to 7 days after the 2nd study vaccination. As pre-specified, data are presented pooled per treatment received for participants in Phases 1/2/3a/3b only.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 8492 | 7940
Participants | 2 | 43

15. Secondary Outcome: Number of Participants With Death Due to COVID-19
Description: Number of participants with death due to COVID-19 in participants with no evidence of prior infection.
Time Frame: Day 36 to Day 92
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 8492 | 7940
Participants | 1 | 9

16. Secondary Outcome: Number of Participants With a First Occurrence of COVID-19 Irrespective of Prior Infection
Description: Number of participants with a first occurrence of COVID-19 irrespective of prior infection.
Time Frame: Day 36 to Day 92
Population: Modified Intent-to-Treat (mITT) Analysis Set (pooled for Phases 1/2/3a/3b), including participants who received both doses of study vaccine and no infection between Day 1 and Day 35 but including those who were seropositive at baseline (Day 1). As pre-specified, data are presented pooled per treatment received for participants in Phases 1/2/3a/3b only.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 8492 | 7941
Participants | 223 | 457

17. Secondary Outcome: Number of Participants With a First Occurrence of COVID-19
Description: Number of participants with a first occurrence of COVID-19 in participants with no evidence of prior infection.
Time Frame: Day 1 to Day 92
Population: Intent-to-Treat (ITT) Analysis Set, which included all participants who received any dose of study vaccine. Participants were analyzed according to the vaccine to which the participant was randomly assigned. As pre-specified, data are presented for participants in the Phase 3b ITT.
Measure: Count of Participants; unit: Participants
Arm/Group | ARCT-154 | Placebo
Number analyzed (Participants) | 8056 | 8044
Participants | 223 | 496

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events (AEs): Day 1 to Day 92, and Day 92 to End of Study (up to approximately Day 394). Other (non-serious) AEs for Phases 1, 2, 3a and 3b: Day 1 to Day 92, and Day 92 to End of Study (up to approximately Day 394) and other (non-serious) AEs for Phase 3c: Day 1-57.
Description: Safety Analysis Set: participants who received vaccine with evaluable data. As pre-specified, data were collected/reported pooled per treatment for Day 1-92&Day 92-End of Study (EOS) for mortality&SAEs. As pre-specified, other AEs for Phases 1,2,3a,3b were collected/reported for Day 1-92 &Day 92-EOS and for Phase 3c Day 1-57. The different data collection periods are reported as distinct arms. AE data were not collected per actual intervention for switchover and re-randomization for 1/2/3a/3b.
Groups:
- Phases 1, 2, 3a, 3b: ARCT-154 Day 1-92: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series (Day 1 and Day 29) of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data for Day 1-92 in this arm are presented for participants who initially received ARCT-154 in Phases 1, 2, 3a, 3b (pooled).
- Phases 1, 2, 3a, 3b: Placebo Day 1-92: This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 micrograms (µg) or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data for Day 1-92 in this arm are presented for participants who initially received placebo in Phases 1, 2, 3a, 3b (pooled).
- Phases 1, 2, 3a, 3b: Placebo or ARCT-154 Day 92-End of Study (Day 394): This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 µg or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series (Day 1 and Day 29) of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data for Day 92- End of Study (Day 394) in this arm are presented for participants who initially received ARCT-154 in Phases 1, 2, 3a, 3b (pooled), and then placebo or ARCT-154 from Day 92-EOS.
- Phases 1, 2, 3a, 3b: ARCT-154 Day 92-End of Study (Day 394): This study was conducted in 3 phases (Phase 1, 2, 3a, 3b, 3c). Phase 1, 2, 3a, 3b: Participants were randomly assigned to receive up to 2 vaccination series at 28-day intervals: an initial vaccination series with vaccinations on Day 1 and Day 29 and an additional vaccination series on Day 92 and 120. Each participant received a two-dose vaccination series of ARCT-154 at a dose of 5 micrograms (µg) or a two-dose vaccination series of placebo (saline) in the first series. In the second vaccination series, participants in Phase 1 and 3b received a two-dose vaccination series with the opposite vaccine on Day 92 and 120 ("Switchover" vaccination series). Participants in Phase 2 and 3a who received 2 doses of ARCT-154 vaccine in the first vaccine series were re-randomized to receive either dose 3 of ARCT-154 on Day 92 plus placebo on Day 120 or placebo on Day 92 plus placebo on Day 120. Phase 3c: Participants were randomly assigned to a study group to receive two-dose vaccination series of ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]). In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data for Day 92- End of Study (Day 394) in this arm are presented for participants who initially received placebo in Phases 1, 2, 3a, 3b (pooled) and then ARCT-154 from Day 92-EOS.
- Phase 3c: ARCT-154 Day 1-92: Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover). As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for ARCT-154 received in Phase 3c from Day 1-92.
- Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-92: Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]) on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for Astra Zeneca COVID-19 vaccine received in Phase 3c from Day 1-92.
- Phase 3c: ARCT-154 Day 92- End of Study (Day 394): Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover). As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for ARCT-154 received in Phase 3c from Day 92- End of Study (Day 394).
- Phase 3c: Astra Zeneca COVID-19 vaccine Day 92-End of Study (Day 394): Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]) on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for Astra Zeneca COVID-19 vaccine received in Phase 3c from Day 92- End of Study (Day 394).
- Phase 3c: ARCT-154 Day 1-57: Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover). As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for ARCT-154 received in Phase 3c from Day 1-57.
- Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-57: Phase 3c: Participants were randomly assigned to a study group to receive ARCT-154 at a dose of 5 µg or approved COVID-19 vaccine comparator (Astra Zeneca's COVID-19 vaccine [ChAdOx1 nCoV-19]) on Day 1 and Day 29. In Phase 3c, participants received only 2 doses of their assigned treatment (no switchover) on Days 1 and 29. As pre-specified, data are presented pooled per treatment received. Data in this arm are presented pooled for Astra Zeneca COVID-19 vaccine received in Phase 3c from Day 1-57.
Arm/Group | Phases 1, 2, 3a, 3b: ARCT-154 Day 1-92 | Phases 1, 2, 3a, 3b: Placebo Day 1-92 | Phases 1, 2, 3a, 3b: Placebo or ARCT-154 Day 92-End of Study (Day 394) | Phases 1, 2, 3a, 3b: ARCT-154 Day 92-End of Study (Day 394) | Phase 3c: ARCT-154 Day 1-92 | Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-92 | Phase 3c: ARCT-154 Day 92- End of Study (Day 394) | Phase 3c: Astra Zeneca COVID-19 vaccine Day 92-End of Study (Day 394) | Phase 3c: ARCT-154 Day 1-57 | Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-57
All-Cause Mortality (participants affected / at risk) | 5/8807 | 16/8294 | 12/8161 | 9/7582 | 0/1186 | 1/1180 | 0/1171 | 3/1168 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 133/8807 | 217/8294 | 180/8161 | 176/7582 | 22/1186 | 35/1180 | 64/1171 | 53/1168 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1303/8807 | 1489/8294 | 1618/8161 | 1374/7582 | 0/0 | 0/0 | 0/0 | 0/0 | 339/1186 | 304/1180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phases 1, 2, 3a, 3b: ARCT-154 Day 1-92 (N=8807) | Phases 1, 2, 3a, 3b: Placebo Day 1-92 (N=8294) | Phases 1, 2, 3a, 3b: Placebo or ARCT-154 Day 92-End of Study (Day 394) (N=8161) | Phases 1, 2, 3a, 3b: ARCT-154 Day 92-End of Study (Day 394) (N=7582) | Phase 3c: ARCT-154 Day 1-92 (N=1186) | Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-92 (N=1180) | Phase 3c: ARCT-154 Day 92- End of Study (Day 394) (N=1171) | Phase 3c: Astra Zeneca COVID-19 vaccine Day 92-End of Study (Day 394) (N=1168) | Phase 3c: ARCT-154 Day 1-57 (N=0) | Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-57 (N=0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | NA | NA
Arrhythmia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | NA | NA
Vertigo positional (Ear and labyrinth disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA
Vestibular disorder (Ear and labyrinth disorders) | 3 | 5 | 11 | 9 | 0 | 4 | 2 | 2 | NA | NA
Angle closure glaucoma (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Cataract (Eye disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | NA | NA
Pterygium (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | NA
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 3 | 1 | NA | NA
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Gastritis (Gastrointestinal disorders) | 2 | 6 | 4 | 2 | 0 | 0 | 0 | 0 | NA | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | NA | NA
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 1 | 5 | 1 | 0 | 0 | 0 | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 5 | 0 | 0 | 0 | 1 | 0 | NA | NA
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA
Type IV hypersensitivity reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Appendicitis (Infections and infestations) | 4 | 2 | 6 | 8 | 0 | 1 | 0 | 2 | NA | NA
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Bronchitis (Infections and infestations) | 0 | 2 | 4 | 2 | 0 | 0 | 2 | 3 | NA | NA
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA
COVID-19 (Infections and infestations) | 50 | 139 | 13 | 17 | 5 | 8 | 4 | 1 | NA | NA
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | NA | NA
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Dengue fever (Infections and infestations) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | NA | NA
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Gastritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | NA | NA
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Peritonitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA
Pneumonia (Infections and infestations) | 2 | 5 | 5 | 5 | 0 | 0 | 4 | 7 | NA | NA
Pneumonia acinetobacter (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Sebaceous gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Septic shock (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | NA | NA
Administration related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | NA | NA
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Foreign body in throat (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2 | 0 | 1 | 1 | 1 | NA | NA
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Spondylopathy traumatic (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | NA | NA
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | NA | NA
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | NA | NA
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | NA | NA
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | NA | NA
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | NA | NA
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Cerebral infarction (Nervous system disorders) | 3 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | NA | NA
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 3 | 2 | 0 | 0 | 2 | 1 | NA | NA
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | NA | NA
Facial paresis (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | NA | NA
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Bipolar I disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 3 | NA | NA
Renal colic (Renal and urinary disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | NA | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA
Genital prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Surgery (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Hypertension (Vascular disorders) | 2 | 0 | 2 | 2 | 1 | 0 | 0 | 2 | NA | NA
Hypertensive crisis (Vascular disorders) | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | NA | NA
Thyroglossal cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA
Allergy to chemicals (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | NA | NA
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA
Snake bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | NA | NA
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 2 | NA | NA
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | NA | NA
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Conductive deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | NA | NA
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | NA | NA
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA
Abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | NA | NA
Bone tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Diabetic foot infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Laryngopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | NA | NA
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | NA | NA
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | NA | NA
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | NA | NA
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 3 | NA | NA
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 0 | NA | NA
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parathyroid disorder (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary gland mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Accidental death (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Necrosis (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dengue haemorrhagic fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body in mouth (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury corneal (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arachnoid cyst (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anembryonic gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Risk of future pregnancy miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephritic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phases 1, 2, 3a, 3b: ARCT-154 Day 1-92 (N=8807) | Phases 1, 2, 3a, 3b: Placebo Day 1-92 (N=8294) | Phases 1, 2, 3a, 3b: Placebo or ARCT-154 Day 92-End of Study (Day 394) (N=8161) | Phases 1, 2, 3a, 3b: ARCT-154 Day 92-End of Study (Day 394) (N=7582) | Phase 3c: ARCT-154 Day 1-92 (N=0) | Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-92 (N=0) | Phase 3c: ARCT-154 Day 92- End of Study (Day 394) (N=0) | Phase 3c: Astra Zeneca COVID-19 vaccine Day 92-End of Study (Day 394) (N=0) | Phase 3c: ARCT-154 Day 1-57 (N=1186) | Phase 3c: Astra Zeneca COVID-19 vaccine Day 1-57 (N=1180)
Tachycardia (Cardiac disorders) | 113 | 96 | 128 | 107 | NA | NA | NA | NA | 0 | 0
COVID-19 (Infections and infestations) | 56 | 123 | 1199 | 1006 | NA | NA | NA | NA | 6 | 14
Influenza (Infections and infestations) | 201 | 188 | 0 | 0 | NA | NA | NA | NA | 83 | 67
Pharyngitis (Infections and infestations) | 106 | 110 | 0 | 0 | NA | NA | NA | NA | 29 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 125 | 132 | 0 | 0 | NA | NA | NA | NA | 34 | 24
Headache (Nervous system disorders) | 281 | 285 | 0 | 0 | NA | NA | NA | NA | 55 | 70
Cough (Respiratory, thoracic and mediastinal disorders) | 128 | 141 | 0 | 0 | NA | NA | NA | NA | 17 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 67 | 91 | 0 | 0 | NA | NA | NA | NA | 0 | 0
Hypertension (Vascular disorders) | 349 | 323 | 291 | 261 | NA | NA | NA | NA | 78 | 60
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | NA | NA | NA | NA | 10 | 15
Fatigue (General disorders) | 0 | 0 | 0 | 0 | NA | NA | NA | NA | 18 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | NA | NA | NA | NA | 12 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | NA | NA | NA | NA | 13 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT05012943/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT05012943/SAP_001.pdf